CLINICAL TRIAL: NCT03982303
Title: A Dose Escalation Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Antitumor Efficacy of Hemay102 in Patients With Advanced Solid Tumors
Brief Title: Phase I Study of Hemay102 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Hemay Oncology Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HM102ST1S01
Record Dates: First submitted 2019-06-09; First posted 2019-06-11 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Patients With Advanced Stage Solid Tumors

STUDY DESIGN:
Masking Description: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Hemay102 at the dosage of 5mg/m2 (Experimental): Hemay102 will be administered to patients through i.v. drip for 4hrs at the dosage of 5mg/m2.
  Interventions: Drug: Hemay102
- Hemay102 at the dosage of 10mg/m2 (Experimental): Hemay102 will be administered to patients through i.v. drip for 4hrs at the dosage of 10mg/m2.
  Interventions: Drug: Hemay102
- Hemay102 at the dosage of 20mg/m2 (Experimental): Hemay102 will be administered to patients through i.v. drip for 4hrs at the dosage of 20mg/m2.
  Interventions: Drug: Hemay102
- Hemay102 at the dosage of 40mg/m2 (Experimental): Hemay102 will be administered to patients through i.v. drip for 4hrs at the dosage of 40mg/m2.
  Interventions: Drug: Hemay102
- Hemay102 at the dosage of 60mg/m2 (Experimental): Hemay102 will be administered to patients through i.v. drip for 4hrs at the dosage of 60mg/m2.
  Interventions: Drug: Hemay102
- Hemay102 at the dosage of 90mg/m2 (Experimental): Hemay102 will be administered to patients through i.v. drip for 4hrs at the dosage of 90mg/m2.
  Interventions: Drug: Hemay102
- Hemay102 at the dosage of 120mg/m2 (Experimental): Hemay102 will be administered to patients through i.v. drip for 4hrs at the dosage of 120mg/m2.
  Interventions: Drug: Hemay102

INTERVENTIONS:
Drug: Hemay102 — Hemay102 was administered through i.v. infusion for 4hrs.

SUMMARY:
This trial was a single-center, open-label, dose-increasing Phase I clinical study with subjects enrolled in patients with advanced solid tumors who failed standard treatment or who were unable to receive effective treatment. The trial is divided into two stages: dose escalation and dose extension.

DETAILED DESCRIPTION:
Dose escalation:

A total of 7 dosage groups were set at this stage, which were 5 mg/m2, 10 mg/m2, 20 mg/m2, 40 mg/m2, 60 mg/m2, 90 mg/m2, and 120 mg/m2, respectively. Accelerated dosage titration was performed in the first 3 dose groups, 1 subject was enrolled in each group; the last 4 dose groups were perfromed into dosage groups by the principle of "3+3" dose increment rule, and the number of subjects enrolled in each group is 3 to 6 cases.

Dose extension:

According to the test results of the dose escalation phase, two extensions of MTD (tentative 60 mg/m2, 90 mg/m2) were selected for the expansion trial. Each dose level was planned to enroll 6 subjects (12 in total), subjects were administered once every 3 weeks (1 treatment cycle every 3 weeks), and received 4 treatment cycles in a row for Hemay102. Safety, tolerability, pharmacokinetic characteristics, and initial anti-tumor efficacy were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and ≤70 years old, male or female;
* A patient who has been confirmed by histology or cytology to have advanced or metastatic solid tumors (in the patients with locally advanced hepatocellular carcinoma or metastatic liver cancer, patients can be recruited by clinical diagnosis) and who have failed standard treatment or who are unable to receive/do not have effective treatment;
* At least one evaluable tumor lesion (spiral CT scan with a long diameter ≥ 10 mm, in accordance with RECIST version 1.1);
* ECOG PS score 0~1 within 1 week before enrollment;
* Estimated survival time of more than 3 months;
* Appropriate hematopoietic function: white blood cell count ≥ 3 × 10^9 / L; absolute neutrophil count ≥ 1.5 × 10^9 / L; platelet count ≥ 100 × 10^9 / L; hemoglobin ≥ 90 g / L;
* Appropriate liver function: total bilirubin ≤ 1.5 × upper limit of normal (ULN); aspartate transferase (AST) ≤ 2.5 × ULN; alanine aminotransferase (ALT) ≤ 2.5 × ULN;
* Proper renal function: serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL / min according to the Cockcroft-Gault formula;
* For clinically confirmed unresectable locally advanced hepatocellular carcinoma or metastatic liver cancer, the patient's liver function must meet the criteria below: ALT≤2.5×ULN, AST≤2.5×ULN, TBIL≤1.5×ULN, Child-Pugh score A or B Grade (≤7 points), blood ammonia ≤100μmol/L (only for patients with hepatocellular carcinoma);
* A qualified male or female patient with fertility must agree to use a reliable method of contraception (hormone or barrier method) after signing the informed consent until at least 12 weeks after the last dose;
* Subjects must give informed consent to the study prior to the trial and voluntarily sign a written informed consent form;
* Subjects are able to communicate well with the investigator and are able to complete the study in accordance with the trial regulations.

Exclusion Criteria:

* Subjects known to have or suspected to have brain metastases;
* Have received radiation therapy within 4 weeks before enrollment;
* Drugs that may affect the metabolism of this product, such as CYP3A4 strong inducer (rifampicin, carbamazepine, phenytoin, etc.) or strong inhibitors (clarithromycin, protease, triazole antifungals, etc.), should be combined within 2 weeks before the study or during the study period;
* Patients who have previously received anthracycline treatment; or who are known to have a history of allergies to anthracyclines (eg, doxorubicin, epirubicin);
* Have active infection or HIV-positive infection or other serious illness;
* Untreated active hepatitis C (anti-HCV antibody positive and HCV RNA positive patients cannot be enrolled); untreated active hepatitis B (HBsAg positive and HBV DNA ≥ 2000 IU/mL) (Note: Hepatitis B subjects treated with treatment also met the inclusion criteria if the following criteria were met: HBV viral load was less than 2000 IU/mL before the first dose of study drug, or patients who are on HBV treatment, and patients with viral load lower than 2000 IU/mL can also be enrolled);
* Uncontrolled or important cardiovascular disease, which included a) New York Heart Association (NYHA) grade II or higher congestive heart failure, unstable angina, myocardial infarction, or arrhythmia requiring treatment (including atrial fibrillation, at screening) within 6 months prior to the first study drug administration Supraventricular tachycardia, ventricular tachycardia or ventricular fibrillation, or left ventricular ejection fraction (LVEF) < 50%; b) Primary cardiomyopathy (eg dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, undetermined cardiomyopathy); c) Clinically significant QTc interval prolongation history, or screening period QTc interval (corrected by Bazette) ≥ 450ms (male) or ≥ 470ms (female); d) Coronary heart disease with symptoms requiring medication; e) Uncontrollable hypertension (refers to post-treatment systolic blood pressure > 160 mmHg and / or diastolic blood pressure > 100 mmHg);
* A history of hemorrhagic or thromboembolic events in the past 6 months, such as cerebrovascular accidents (including transient ischemic attacks), pulmonary embolism, and spontaneous bleeding of the tumor;
* Medical treatment for other clinical trials within 4 weeks prior to enrollment;
* <4 weeks after major surgery or trauma after enrollment;
* Must take other treatments during the trial, such as other chemotherapy, targeted therapy, hormone therapy, immunotherapy, radiotherapy (except for local symptomatic radiotherapy) or Chinese medicine;
* Concomitant mental illness;
* The investigator believes that the subject is not suitable for this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | from baseline until 4 weeks after the study day
  Number of participants with adverse events

SECONDARY OUTCOMES:
Objective response rate | At screening, every 6 weeks of treatment up to 18 months
  Objective response rate (complete response rate + partial response rate) according to RECIST v1.1
Clinical benefit rate | At screening, every 6 weeks of treatment up to 18 months
  Clinical benefit rate defined as percentage of patients with stable disease (SD) ≥ 6 months/partial response (PR)/complete response (CR). according to RECIST v1.1
Progression Free Survival | 18 months after treatment initiation
  Progression Free Survival defined as the proportion of patients alive and without progression (according to RECIST v1.1 criteria)
AUC | 0, 1, 2, 3, 5, 8, 12, 24, 48 and 72 hours post-dose
  Area under the plasma concentration versus time curve of Hemay102

CONTACTS AND LOCATIONS:
Overall Officials: Ti Zhang, Ph.D., Principal Investigator — Tianjing medical university cancer hospital
Locations (1):
- Tianjin medical university cancer hoapital, Tianjin, China